CLINICAL TRIAL: NCT03117686
Title: Estimation of Pulmonary Arterial Pressure With Transesophageal Echocardiography: A Pilot Study
Brief Title: Lung Ultrasound in High Altitude Lung Edema
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ulrike Weber, Ass.Prof.Dr., Medical University of Vienna
Other Study IDs: 1236/2017
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Edema
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: 10 healthy volunteers climbing Mount Kilimanjaro receiving lung ultrasound
  Interventions: Diagnostic Test: lung ultrasound
- patients after lung transplantation: 10 patients > 2years after lung transplantation climbing Mount Kilimanjaro receiving lung ultrasound
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — lung ultrasound with positive "B-line pattern" in patients after lung transplantations and healthy volunteers at sea level and high altitude (4600 m) at Mountb Kilimanjaro

SUMMARY:
High altitude pulmonary edema is a life-threatening condition that remains a concern for climbers and clinicians alike. It is defined as a non-cardiac pulmonary edema occurring at altitudes exceeding 3000m in non-acclimatised individuals. Recently, studies conducted in remote areas have demonstrated that ultrasound lung comets (B lines) can be used as a measure of sub-acute pulmonary edema and high altitude pulmonary edema in climbers ascending to altitude. the investigators want to assess the occurrence of of comet tails (B lines) as a measure of pulmonary edema among patients after lung transplantation and healthy individuals during an expedition to Mount Kilimanjaro.

DETAILED DESCRIPTION:
High altitude pulmonary edema is a life-threatening condition that remains a concern for climbers and clinicians alike. It is defined as a non-cardiac pulmonary edema occurring at altitudes exceeding 3000m in non-acclimatised individuals. Within the last decade, studies have shown ultrasonography to be valuable in the accurate diagnosis of a variety of lung pathologies, including cardiogenic pulmonary edema, pleural effusion, pneumothorax, and lung consolidation. Recently, studies conducted in remote areas have demonstrated that ultrasound lung comets (B lines) can be used as a measure of sub-acute pulmonary edema and high altitude pulmonary edema in climbers ascending to altitude. These studies also demonstrated that small portable ultrasound devices are reliable at high altitude in a cold and hypobaric environment.

So far all studies concerning the detection of comet tails as a measure of pulmonary edema have been done only in a healthy population. There is no study evaluating this topic in patients after lung transplantation.

Study objectives (Hypothesis)

The investigators want to assess the occurrence of of comet tails (B lines) as a measure of pulmonary edema among patients after lung transplantation and healthy individuals during an expedition to Mount Kilimanjaro.

Study design

Prospective observational single-center study.

Study population

10 patients > 2 years after lung transplantation and 10 healthy volunteers

Methods

The investigators will do the ultrasound examinations using the portable V-scan ultrasonography device (GE Healthcare) with a dual probe, including a phased array cardiac probe on one side and a linear probe on the other side.

Examinations will be done at sea level (before and right after the expedition), on the 3rd day at Shira hut at 3840 m and on the 6th day at Barafu camp at 4600m (highest camp site before summiting). Examinations will be done at the camp sites in a tent to assure good examination conditions for the patients.

Lung ultrasound will be performed with the patient in supine position. The phased-array transducer will be used for lung ultrasound, and will be used for the assessment of B-lines, which arise from the pleural line to the bottom of the screen and move with the sliding lung. The investigators will quantify the B- line burden in lung regions using the validated Eight-region method: Each hemithorax is divided into four quadrants, upper and lower anterior and upper and lower lateral divided longitudinally by the anterior axillary line and transversely by the 2nd intercostal space. If 3 or more B-lines (any size and spaced apart by any distance) are present in a particular region, that region is considered positive. Two or more positive regions per side define a "B-line pattern."

Measurement of optic nerve sheath diameter will be performed with a linear transducer placed superior and lateral to the eye, above the upper eyelid. The patient will be positioned supine, with a 30 degree head elevation. After visualization of the entry of the optic nerve into the globe, we will freeze the image. Optic nerve sheath diameter will be measured 3mm behind the globe in a perpendicular axis to the nerve. Two measurements will be taken per eye, and the mean of the 4 values will represent the optic nerve sheath diameter. A nerve sheath diameter of more than 5.8mm is defined as equivalent with an intracranial pressure (ICP) of more than 20mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Expedition to Mount Kilimanjaro

Exclusion Criteria:

* Refusal to participate in the study
* Age < 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 patients > 2 years after lung transplantation and 10 healthy volunteers during expedition to Mount Kilimanjaro
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
lung ultrasound | 2 weeks
  Positive "B-line pattern" in patients after lung transplantations and healthy volunteers at sea level and high altitude (4600 m)

SECONDARY OUTCOMES:
optic nerve sheath diameter | 2 weeks
  optic nerve sheath diameter in patients after lung transplantations and healthy volunteers at sea level and high altitude (4600 m)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Weber, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical university of vienna, General hospital of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No